CLINICAL TRIAL: NCT03726320
Title: Randomized Trial of Community Health Worker-led Decision Coaching to Promote Shared Decision Making for Prostate Cancer Screening Among Black Male Patients and Their Providers
Brief Title: Trial of Community Health Worker-led Decision Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 18-00514; 1R01MD012243-01A1 (NIH)
Record Dates: First submitted 2018-09-07; First posted 2018-10-31 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A decision aid along with decision coaching on PSA screening from a Community Health Worker (CHW). The intervention will be administered directly prior to the participant's appointment with their provider.
  Interventions: Behavioral: Education Counseling Session for PSA Screening
- Control Group (Active Comparator): A decision aid along with CHW interaction on dietary and lifestyle modification to serve as an attention control. The intervention will be administered directly prior to the participant's appointment with their provider.
  Interventions: Behavioral: General Health Counseling Coaching

INTERVENTIONS:
Behavioral: Education Counseling Session for PSA Screening — counseling from extensively trained CHW
  Arms: Intervention Group
Behavioral: General Health Counseling Coaching — coaching using an educational tool focused on dietary and lifestyle modification
  Arms: Control Group

SUMMARY:
Black men are disproportionately affected by prostate cancer, the most common non-cutaneous malignancy among men in the U.S. This randomized trial will evaluate the efficacy of a Community Health Worker-led decision coaching program to facilitate Shared Decision Making (SDM) and Prostate Specific Antigen (PSA) screening among Black men with regards to decision quality, the decision making process, patient-provider communication and PSA utilization for Black men in the primary care setting.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Black
* Male
* Attending FQHC for routine primary care appointment

Providers:

* Provider at Sunset Park Health Council Federally Qualified Health Center (FQHC)
* Caring for patients that fit inclusion criteria

Exclusion Criteria:

* Provider at Sunset Park Health Council Federally Qualified Health Center (FQHC)
* Caring for patients that fit inclusion criteria

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender Identity
Enrollment: 162 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danil Makarov, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided).Researchers who provide a methodologically sound proposal will have access to the data.

REFERENCES:
- [Derived] Makarov DV, Feuer Z, Ciprut S, Lopez NM, Fagerlin A, Shedlin M, Gold HT, Li H, Lynch G, Warren R, Ubel P, Ravenell JE. Randomized trial of community health worker-led decision coaching to promote shared decision-making for prostate cancer screening among Black male patients and their providers. Trials. 2021 Feb 10;22(1):128. doi: 10.1186/s13063-021-05064-4. PMID 33568208

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in the Patient Providers arm were not assigned to an intervention/control condition. Rather, these providers treated patient participants assigned to both the intervention group and the control group. As such, Participant Flow data on the Patient Provider participants is presented in 1 arm.
Groups:
- Intervention Group: Patients: A decision aid along with decision coaching on PSA screening from a Community Health Worker (CHW). The intervention will be administered directly prior to the participant's appointment with their provider.
  Education Counseling Session for PSA Screening: counseling from extensively trained CHW
- Control Group: Patients: A decision aid along with CHW interaction on dietary and lifestyle modification to serve as an attention control. The intervention will be administered directly prior to the participant's appointment with their provider.
  General Health Counseling Coaching: coaching using an educational tool focused on dietary and lifestyle modification
- Patient Providers: Patient provider participants included patients' physicians/nurse practitioners. Patient provider participants had appointments with both control and intervention patients.
Period: Overall Study
Arm/Group | Intervention Group: Patients | Control Group: Patients | Patient Providers
Started | 66 | 68 | 12
Completed | 54 | 60 | 11
Not Completed | 12 | 8 | 1
Not completed — Lost to Follow-up | 2 | 4 | 0
Not completed — Time Constraints | 4 | 1 | 0
Not completed — Ineligible after enrollment | 3 | 3 | 0
Not completed — Clinic / insurance issue | 2 | 0 | 0
Not completed — Language barrier | 1 | 0 | 0
Not completed — Provider left the clinic | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Patient Providers: Patient provider participants included patients' physicians/nurse practitioners.
- Total: Total of all reporting groups
Arm/Group | Intervention Group: Patients | Control Group: Patients | Patient Providers | Total
Number analyzed (Participants) | 54 | 60 | 12 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (8.72) | 54.7 (7.63) | 41.7 (10.1) | 49.87 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex information is missing from 1 participant in the patient provider arm.
  Participants
    number analyzed (Participants) | 54 | 60 | 11 | 125
    Female | 0 | 0 | 8 | 8
    Male | 54 | 60 | 3 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 0 | 0 | 10 | 10
  Unknown or Not Reported | 54 | 59 | 0 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 54 | 60 | 4 | 118
  White | 0 | 0 | 3 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 54 | 60 | 12 | 126

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Screening Rates
Description: Percentage of participants who receive at least one PSA screening. Screening data are collected through patient self-reports and electronic health record data.
Time Frame: Up to Month 3
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
Percentage of participants | 77.8 | 76.7

2. Primary Outcome: Patient Knowledge Survey Score
Description: The Patient Knowledge Survey comprises 12 items assessing participants' understanding of PSA testing and prostate cancer. Respondents provide an answer of "True," "Unsure," or "False." The total score is the sum of correct responses and ranges from 0-12; higher scores indicate greater knowledge.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
score on a scale | 8.13 (1.33) | 5.23 (2.24)

3. Primary Outcome: Decision Quality Score
Description: Scale consists of 12 items assessing participants' attitudes toward prostate cancer treatment and screening (6 Pros and 6 Cons of testing) scored on a 5 point Likert scale (Strongly Disagree to Strongly Agree). The total score is the sum of responses and ranges from -24 to +24; Positive scores indicate a more favorable assessment of the pros versus the cons of the test.This survey will be administered twice: once directly following the coaching session prior to the patient's appointment, and again following the appointment.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
score on a scale | 11.2 (5.42) | 10.8 (3.99)

4. Primary Outcome: Percentage of Participants Who Make Informed Choice
Description: Percentage of participants who made an Informed Choice to either undergo or decline PSA testing. Informed choices are those in which:
  1. Men with good knowledge and positive measure of informed choice attitudes (> or = 22) choose to undergo the test OR 2) Men with good knowledge but negative measure of informed choice attitudes (<22) towards the test, do not undergo the test The Measure of Informed Choice Attitudes survey is administered twice: once directly following the coaching session prior to the patient's appointment, and again following the appointment and the patient's screening decision is recorded during post-appointment.
Time Frame: Day 1
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
Percentage of participants | 64.8 | 43.3

5. Secondary Outcome: Decision Self-Efficacy Scale Score
Description: The Decision Self-Efficacy Scale is an 11-item survey measuring confidence in making an informed choice. Each item is rated on a scale from 0-4, where 0 = not at all confident and 4 = very confident. The raw score is the sum of responses and is transformed to a standard total score ranging from 0 to 100; higher scores indicate "extremely high self-efficacy."
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
score on a scale | 96 (8.41) | 94.7 (9.15)

6. Secondary Outcome: Doctor-Patient Communication Survey Score
Description: The Doctor-Patient Communication Survey includes 19 items assessing how participants felt they were able to communicate with their provider. Each item is rated on a scale from 1-5, where 1 = strongly disagree and 5 = strongly agree. The total score is the average score of responses and ranges from 0 to 5; higher scores indicate greater doctor-patient communication.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
score on a scale | 4.28 (0.395) | 4.31 (0.412)

7. Secondary Outcome: Perceived Efficacy in Patient-Physician Interactions Questionnaire (PEPPI) Score
Description: PEPPI is a 10-item assessment of participant's perceived self-efficacy for communicating with their provider. Each item is rated on a scale from 1-5, where 1 = not at all confident and 5 = very confident. The total score is the sum of responses and ranges from 10 to 50; higher scores indicate greater self-efficacy in communicating with providers.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
score on a scale | 47.5 (4.86) | 47.3 (4.4)

8. Secondary Outcome: Change in Decisional Conflict Scale Score
Description: The Decisional Conflict Scale is a 16-item survey assessing the level of decisional conflict for participants when deciding whether to have prostate cancer screening. Each item is rated on a 0-4 scale, where 0 = strongly agree and 4 = strongly disagree. The total score is the sum of responses and ranges from 0 to 64. Scores lower than 25 are associated with implementing decisions; scores exceeding 37.5 are associated with decision delay or feeling unsure about implementation.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
score on a scale | 17 (11) | 21.9 (13.2)

9. Secondary Outcome: Satisfaction With Decision Scale Score
Description: 6-item assessment of participants' satisfaction with their prostate cancer screening decisions. Each item is rated on a 1-5 scale, where 1 = strongly disagree and 5 = strongly agree. The total score is the average of all items and ranges from 1-5. Higher scores indicate greater satisfaction with decision.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 54 | 60
score on a scale | 4.48 (0.48) | 4.31 (0.539)

10. Secondary Outcome: Decisional Regret Scale Survey
Description: 5-item assessment of participants' regret toward the first decision they made about prostate cancer screening after speaking with their provider. Each item is rated on a scale from 1-5, where 1 = strongly agree and 5 = strongly disagree. The total score is the sum of responses and ranges from 5 to 25. Higher scores indicate greater regret. To help others interpret the score more readily with other scales ranging from 0 to 100, these scores can then be converted to a 0-100 scale by subtracting 1 from each item then multiply by 25. To obtain a final score, the items are summed and averaged. The final score presented ranges from 0 to 100, higher scores indicate greater regret.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 51 | 49
score on a scale | 21.2 (15.3) | 27 (18.2)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The occurrence of an AE or SAE may come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care, or upon review by a study monitor. Note that participants in the patient provider arm were not assessed for deaths or adverse events.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/60
Other Adverse Events (participants affected / at risk) | 0/54 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03726320/Prot_SAP_000.pdf